CLINICAL TRIAL: NCT00480207
Title: Randomized Double-blind Controlled Clinical Trial to Assess the Impact of Folic Acid and Omega-3 Fatty Acids Supplementation on the Severity of Depressive Symptoms in Older Adults With Identified Depression
Brief Title: Folic Acid and Omega -3 Fatty Acid Supplementation in Depressed Older Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Prof. RH Belmaker (Other Government)
Collaborators: The S. Daniel Abraham International Center for Health and Nutrition (Other)
Responsible Party: Sponsor-Investigator, Prof. RH Belmaker, Prof. RH Belmaker, Beersheva Mental Health Center
Organization: Beersheva Mental Health Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ICHN-4413
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Folic Acid; Docosahexaenoic Acids; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- omega-3, folic acid, vitB12 (Experimental): folic acid (1600 mcg per day), and omega-3 (2000 mg per day: active docosahexaenoic acid (DHA) and eicosapentanoic acid (EPA), proportion 1:1), vitamin B12 (1000 mcg per day)
  Interventions: Dietary Supplement: folic acid; Dietary Supplement: omega-3; Dietary Supplement: vit B12
- omega-3, folic acid placebo, vit B12 (Experimental): omega-3,folic acid placebo (starch), vitamin B12 (1000 mcg per day)
  Interventions: Dietary Supplement: omega-3; Dietary Supplement: vit B12; Other: folic acid placebo
- omega-3 placebo, folic acid, vit B12 (Experimental): folic acid, omega-3 placebo(canola oil),vitamin B12 (1000 mcg per day)
  Interventions: Dietary Supplement: folic acid; Dietary Supplement: vit B12; Other: omega-3 placebo
- omega-3 placebo, folic acid placebo, vit B12 (Experimental): omega-3 placebo (canola oil),folic acid placebo (starch), vitamin B12 (1000 mcg per day)
  Interventions: Dietary Supplement: vit B12; Other: folic acid placebo; Other: omega-3 placebo

INTERVENTIONS:
Dietary Supplement: folic acid
  Arms: omega-3 placebo, folic acid, vit B12; omega-3, folic acid, vitB12
Dietary Supplement: omega-3
  Arms: omega-3, folic acid placebo, vit B12; omega-3, folic acid, vitB12
Dietary Supplement: vit B12
Other: folic acid placebo
  Arms: omega-3 placebo, folic acid placebo, vit B12; omega-3, folic acid placebo, vit B12
Other: omega-3 placebo
  Arms: omega-3 placebo, folic acid placebo, vit B12; omega-3 placebo, folic acid, vit B12

SUMMARY:
Our specific aim is to determine the impact of folic acid and omega-3 supplementation on the severity of depressive symptoms among depressed adults aged 65 and above.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65+ (year of birth -1942 or below)
2. Depression (as defined by the DSM-IV diagnostic criteria for depression: major or minor depression or dysthymia)

Exclusion Criteria:

1. Co-existing psychiatric disorder (except anxiety disorders)
2. Moderate and severe cognitive impairment
3. Current treatment with anticoagulants, antithrombotics and fibrinolytics
4. Current severe angina with exertion
5. Chronic renal insufficiency
6. Liver cirrhosis
7. Alcohol or drug abuse

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
the severity of depressive symptoms | baseline, 4th , 8th and 12th week

SECONDARY OUTCOMES:
cognitive status | baseline, 4th, 8th, and 12th week
nutritional status | baseline and end of study
possible side effects | baseline, 4th, 8th, and 12th week

CONTACTS AND LOCATIONS:
Overall Officials: Danit R Shahar, RD PhD, Study Director — Ben-Gurion University of the Negev; Alex Palatnik, MD, Principal Investigator — Beersheva Mental Health Center; Larissa German, MD, MMedSc, Principal Investigator — The S. Daniel Abraham International Center for Health and Nutrition
Locations (1):
- Mental Health Center, Beersheba, Israel

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851